CLINICAL TRIAL: NCT03836703
Title: Doubling the Iron Dose VS Single Dose Iron Supplementation to Prevent Iron Deficiency Anemia (IDA) in Twin Pregnant Women: A Randomized Controlled Trial
Brief Title: Doubling the Iron Dose to Prevent IDA in Twin Pregnant Women
Acronym: IDA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Abass, Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3201
Record Dates: First submitted 2019-02-08; First posted 2019-02-11 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Hematologic Pregnancy Complications
Keywords: Pregnancy, Twins , Iron Deficiency Anaemia
MeSH Terms: conditions — Pregnancy Complications, Hematologic; Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single Dose Daily Iron (Active Comparator): single dose daily Iron'IRON FUM&POLYSAC#1/FA/MV NO.18 162 Mg-115.2 Mg (106 Mg Iron)-1 Mg ORAL CAPSULE supplementation From 14 weeks gestation to prevent iron deficiency anemia
  Interventions: Drug: Feroglobin single daily use
- Double dose Daily iron (Experimental): Double dose daily Iron'IRON FUM&POLYSAC#1/FA/MV NO.18 162 Mg-115.2 Mg (106 Mg Iron)-1 Mg ORAL CAPSULE supplementation From 14 weeks gestation to prevent iron deficiency anemia
  Interventions: Drug: Feroglobin twice daily dose

INTERVENTIONS:
Drug: Feroglobin single daily use — Feroglobin single daily use ( IRON FUM&POLYSAC#1/FA/MV NO.18 162 Mg-115.2 Mg (106 Mg Iron)-1 Mg ORAL CAPSULE ) to prevent iron deficiency anemia during pregnancy from 14 weeks gestation going on.
  Other Names: IRON FUM&POLYSAC#1/FA/MV NO.18 162 Mg-115.2 Mg (106 Mg Iron)-1 Mg ORAL CAPSULE
  Arms: Single Dose Daily Iron
Drug: Feroglobin twice daily dose — Feroglobin twice daily dose ( IRON FUM&POLYSAC#1/FA/MV NO.18 162 Mg-115.2 Mg (106 Mg Iron)-1 Mg ORAL CAPSULE ) to prevent iron deficiency anemia during pregnancy from 14 weeks gestation going on.
  Other Names: 'IRON FUM&POLYSAC#1/FA/MV NO.18 162 Mg-115.2 Mg (106 Mg Iron)-1 Mg ORAL CAPSULE
  Arms: Double dose Daily iron

SUMMARY:
In twin pregnancies, the maternal iron demands are magnified, estimated at 1.8 times more than in singleton pregnancies due to greater maternal red blood cell mass and plasma volume expansion as well as increased fetal and placental requirements.

With a lack of randomized controlled trials assessing the adequacy of iron supplements on twin pregnancy, various recommendations are based on level 3 clinical expert opinions at most.

DETAILED DESCRIPTION:
Iron deficiency anemia (IDA) is a very prevalent condition in pregnancy, affecting nearly 18% of all pregnant women during all three trimesters, with as many as 29%of women affected during the third trimester.

In twin pregnancies, the maternal iron demands are magnified, estimated at 1.8 times more than in singleton pregnancies due to greater maternal red blood cell mass and plasma volume expansion as well as increased fetal and placental requirements. Thus, maternal hemoglobin (Hgb) in multiple pregnancies is lower in all trimesters compared with singleton gestations, with a rate of IDA estimated to be 2.4 to even 4 times higher.

Expert opinion relying on the increased risk for micronutrient deficiency in twin pregnancies recommends supplementation of iron beyond that contained in a typical prenatal vitamin. Moreover, some experts support doubling the dose of multivitamins containing 30 mg of elemental iron during the second and third trimesters of a twin pregnancy, regardless of maternal Hgb and ferritin concentrations.

With a lack of randomized controlled trials assessing the adequacy of iron supplements on twin pregnancy, various recommendations are based on level 3 clinical expert opinions at most. The purpose of our study was to assess the efficacy of a single versus a double daily iron supplement dose in iron deficient women with twin pregnancies. Determining the effect of this intervention on maternal iron stores and immediate neonatal outcome measures will assist in defining evidence based recommendations for prenatal care.

ELIGIBILITY:
Inclusion Criteria:

* Twin pregnancy.
* Hemoglobin ≥ 10.5 gm/d l. at booking visit

Exclusion Criteria:

* Continuous hyper-emesis gravid arum lasting beyond 20 weeks of gestation
* Thalassemia minor (alpha or beta).
* Mal-absorption disorders (such as inflammatory bowel diseases, Crohn's disease, ulcerative colitis, previous bowel resection).
* Anemia from chronic illness.
* Any use of multi-vitamin supplements containing iron.
* Any chronic blood loss. e.g: hemorrhoids.
* Autoimmune disorders.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 450 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Hemoglobin level below 11 g/dl | 32 weeks gestation
  Iron deficiency anemia
Hemoglobin level below 11 g/dl | 24 hours before delivery
  incidence of Iron deficiency anemia

SECONDARY OUTCOMES:
blood product administration | 24 hours after delivery
  Number of times of need for blood transfusion at delivery time
GIT side effects | all over the pregnancy time 14 weeks gestation to delivery
  Incidence of Complications of iron supplementation mostly are GIT related
Preterm Birth | delivery before 37 weeks gestation
  number of preterm birth
neonatal Birth weidht | 5 min. after delivery
  birth weight in Kg

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Ibrahem, Prof, Study Chair — AinShams U
Locations (1):
- Ahmed Abass, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shinar S, Skornick-Rapaport A, Maslovitz S. Iron Supplementation in Twin Pregnancy - The Benefit of Doubling the Iron Dose in Iron Deficient Pregnant Women: A Randomized Controlled Trial. Twin Res Hum Genet. 2017 Oct;20(5):419-424. doi: 10.1017/thg.2017.43. Epub 2017 Aug 22. PMID 28829001
- [Background] Tolkien Z, Stecher L, Mander AP, Pereira DI, Powell JJ. Ferrous sulfate supplementation causes significant gastrointestinal side-effects in adults: a systematic review and meta-analysis. PLoS One. 2015 Feb 20;10(2):e0117383. doi: 10.1371/journal.pone.0117383. eCollection 2015. PMID 25700159